CLINICAL TRIAL: NCT03983109
Title: Identify the Epidural Space With EpiFaith Syringe in Air and Saline Based Procedures
Brief Title: EpiFaith Syringe for Epidural Space Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flat Medical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EPS01
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Epidural Localization
Keywords: EpiFaith; Epidural localization

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Detection by EpiFaith syringe with air (Experimental): Fill the EpiFaith Syringe with air for LOR detection
  Interventions: Device: EpiFaith loss of resistance detect syringe
- Detection by EpiFaith syringe with saline (Experimental): Fill the EpiFaith Syringe with saline for LOR detection
  Interventions: Device: EpiFaith loss of resistance detect syringe

INTERVENTIONS:
Device: EpiFaith loss of resistance detect syringe — An EpiFaith syringe will be used to detect the loss of resistance and facilitate the needle localization.

SUMMARY:
The objective of the study is to verify the efficacies of both air and saline based procedure of EpiFaith syringe for assisting the needle localization of the epidural space.

DETAILED DESCRIPTION:
This is a single blind, randomized study. Subjects who will receive a surgery requiring epidural anesthesia or analgesia and meet all of the study criteria will be enrolled in the study. All subjects must sign an informed consent and receive a copy of the signed and dated informed consent form prior to participation in the trial.

The study consists of 2 study visits: Visit 1 (Screening Visit) and Visit 2 (Operative Visit). After screening, eligible subject will be randomly assigned to one of the following groups: Group A: detection by EpiFaith syringe with air; Group S: detection by EpiFaith syringe with saline with a 1:1 ratio. In Visit 2, the following variables will be recorded and rated during the process of epidural space localization: Success of epidural localization, time to identify the epidural space, duration of the epidural space localization procedure, number of attempts, Number of the occurrence of false positive, the distance from the skin to the epidural space, and number of change insertion segment. Adverse events and concomitant treatments will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* Surgery requiring epidural anesthesia or analgesia
* ASA Physical Status 1 to 3

Exclusion Criteria:

* Bleeding and clotting disorders

  * Platelet count < 100,000 / mm3
  * International normalized ratio (INR) > 1.5
* History of peripheral neuropathy
* Neuromuscular or neuropsychiatric disease
* Marked spinal deformities or a history of spinal instrumentation
* Systemic infection
* Skin infection at the injection site
* Significant heart failure, e.g. New York Heart Association (NYHA) Functional Classification 3 or 4

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will be randomized to one of the two groups (A group - EpiFaith syringe with air or S group - EpiFaith syringe with saline) at the ratio of 1:1. The randomization method will result in sealed, opaque envelopes containing the computer- generated, random assignment. Randomization will occur in blocks so that blocks of equal numbers of subjects will be used to avoid potential runs of assignments.
Period: Overall Study
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Started | 30 | 30
Completed | 18 (12 cases were withdrawn because the operator found air pressure cannot be maintained when the operator pushed the plunger to engage the indicator.) | 30
Not Completed | 12 | 0
Not completed — Operational Hurdles Linked to Usage Methodologies | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.83 (10.47) | 61.13 (12.24) | 59.48 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 11 | 17 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.57 (4.31) | 23.82 (3.6) | 24.14 (3.92)
ASA Physical Status [Count of Participants; unit: Participants] — The ASA physical status classification system (October 15, 2014) is a system for assessing the fitness of patients before surgery.
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    Status 1 | 3 | 3 | 6
    Status 2 | 21 | 21 | 42
    Status 3 | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Success of Epidural Localization
Description: Defined as the catheter can be inserted into epidural space successfully, no cold perception in the blocked dermatomes after the injection of anesthetic by cold sensation test, and no occurrence of inadvertent dural puncture.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
Participants
  Success of epidural localization | 18 | 30
  Failure of epidural localization | 0 | 0

2. Secondary Outcome: The Time to Identify the Epidural Space
Description: Defined as the time of the successful localization from the first syringe attached to the Tuohy needle to the occurrence of LOR signal.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
secs | 231 (273) | 130 (169)

3. Secondary Outcome: Duration of the Epidural Space Localization Procedure
Description: Defined as the time from the puncture of skin to the successful insertion of the epidural catheter.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
secs | 309 (276) | 194 (182)

4. Secondary Outcome: Number of Attempts
Description: Defined as the insertion of the epidural catheter is unsuccessful or the perception of cold exists in the blocked dermatomes after the injection of anesthetic by cold sensation test.
Time Frame: 30 minutes
Measure: Median (Full Range); unit: attempts
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
attempts | 2 [1 to 4] | 1 [1 to 4]

5. Secondary Outcome: The Distance From the Skin to the Epidural Space
Description: Defined as the insertion distance of the needle after locating the epidural space.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
mm | 63.3 (10.4) | 65.1 (9.2)

6. Secondary Outcome: Number of Change Insertion Segment
Description: Number of change insertion segment during the epidural localization procedure.
Time Frame: 30 minutes
Measure: Median (Full Range); unit: segments
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
segments | 0 [0 to 1] | 0 [0 to 1]

7. Secondary Outcome: Number of the Occurrence of False Positive
Description: the insertion of the epidural catheter is unsuccessful or the perception of cold exists in the blocked dermatomes after the injection of anesthetic by cold sensation test
Time Frame: 30 minutes
Measure: Median (Full Range); unit: occurrences
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
Number analyzed (Participants) | 18 | 30
occurrences | 0 [0 to 2] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Detection by EpiFaith Syringe With Air | Detection by EpiFaith Syringe With Saline
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT03983109/Prot_SAP_000.pdf